CLINICAL TRIAL: NCT03665337
Title: Reducing Risk: A Comprehensive mHealth Sleep Health Intervention for Adolescents at Risk for Depression and Anxiety Disorders
Brief Title: The Reducing Risk Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-47676
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Insomnia; Delayed Sleep Phase
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are asked to refrain from mentioning any information about the treatment they receive when interacting with the investigator or outcomes assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mTranS-C (Experimental): Access to a mobile and computer accessible adaptation of Transdiagnostic Sleep and Circadian Intervention
  Interventions: Behavioral: mTranS-C
- Control (Active Comparator): Access to a mobile and computer accessible control intervention that targets coping skills and sleep education.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: mTranS-C — MOBILE HEALTH
  Arms: mTranS-C
Behavioral: Control — MOBILE HEALTH
  Arms: Control

SUMMARY:
The present study will test an innovative mobile health adaptation of a behavioral intervention that improves sleep and mental health concerns among adolescents.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* any current psychiatric illness
* currently use of medications or herbs with known effects on sleep
* hospitalization for substance use or suicide within the past 12 months
* known sleep apnea
* unstable major medical conditions
* current psychotherapy for depression, anxiety or sleep health deficits

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | baseline to end of treatment (anticipated average exposure 2 months), months 3 and 8
  Validated questionnaire; total score range between 0 and 21, with higher numbers representing worse sleep quality

SECONDARY OUTCOMES:
Change in the PHQ-9 (The 9 Item Patient Health Questionnaire For Depression) | baseline to end of treatment (anticipated average exposure 2 months), months 3 and 8
  A validated questionnaire measuring depressive symptom severity. The total score ranges between 0 and 19. Scores are rated as minimal (0-4), mild (5-9), moderate (10-14), and severe (15-19).
Change in the SCARED (Screen for Child Anxiety Related Disorders) total score | baseline, and at months 1, 2, 3 and 8
  A validated 41-item questionnaire assessing self-report of anxiety in children and adolescents. Individual items are rated 'Not True or Hardly Ever True' (Score 0), 'Somewhat True or Sometimes True' (Score 1), or 'Very True or Often True' (Score 2). Individual response scores are then summed and for a total score. Total scores range from 0 to 82.
Change in cortisol reactivity and recovery in response to a stress exposure | baseline and at month 3
  A validated biological measure of stress reactivity and recovery in response to a stress exposure. Changes in cortisol production at 15, 30 and 45 minutes following a stressor will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Asarnow, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No